CLINICAL TRIAL: NCT06254014
Title: A Phase 3, Multi-center, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of JY09 in Patients With T2DM Inadequately Controlled by Diet and Exercise Alone
Brief Title: A Phase 3 Study to Evaluate the Efficacy of JY09 Compared With Placebo in T2DM Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFBT-JY09-DM-301
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized in a 1:1:1 ratio to the 1.2 mg JY09 injection group (n=90 cases), the 2.4 mg JY09 injection group (n=90 cases), and the placebo group (n=90 cases).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses a double-blind technique, which means that neither the investigator nor the subject knows what drug is being used. The sponsor will provide the study drug and the control drug, ensuring that the placebo shape, color, and weight are identical to the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exendin-4 Fc fusion protein injection(1.2mg） (Experimental): 1.2mg,Subcutaneous injection in the abdomen,Bi-weekly for 54 weeks.
  Interventions: Drug: Exendin-4 Fc fusion protein injection
- Exendin-4 Fc fusion protein injection(2.4mg） (Experimental): The first dose of 1.2 mg of JY09 injection was administered, the dose was adjusted to 2.4 mg after two weeks, after which 2.4 mg was maintained to continue subcutaneous injection in the abdomen, bi-weekly treatment for 52 weeks.
  Interventions: Drug: Exendin-4 Fc fusion protein injection
- placebo(0.6ml） (Placebo Comparator): JY09 placebo injection 0.6 ml, biweekly abdominal subcutaneous injection for 26 weeks, followed by randomization in a 1:1 ratio into JY09 (1.2 mg) and JY09 (2.4 mg) for 28 weeks, biweekly subcutaneous injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exendin-4 Fc fusion protein injection — 1.2mg, subcutaneous injection in the abdomen, biweekly, 54 weeks of treatment.
  Other Names: JY09(1.2mg)
  Arms: Exendin-4 Fc fusion protein injection(1.2mg）
Drug: Exendin-4 Fc fusion protein injection — The first dose of 1.2 mg was administered subcutaneously in the abdomen, and after two weeks, the dose was adjusted to 2.4 mg, followed by a continuation of treatment for 52 weeks.
  Other Names: JY09(2.4mg)
  Arms: Exendin-4 Fc fusion protein injection(2.4mg）
Drug: Placebo — 0.6 ml, placebo injection, biweekly subcutaneous abdominal injections for 26 weeks (core treatment period), after which placebo was randomized 1:1 to JY09 (1.2 mg) and JY09 (2.4 mg) continued subcutaneous abdominal injections biweekly for 28 weeks (extended treatment period).
  Other Names: Injection mimetic
  Arms: placebo(0.6ml）

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of JY09 versus placebo in patients with type 2 diabetes mellitus (T2DM) inadequately controlled by diet and exercise alone

DETAILED DESCRIPTION:
This study was designed as a multicenter, randomized, double-blind, placebo-parallel controlled Phase III clinical study to evaluate the efficacy and safety of Exendin-4Fc fusion protein (JY09) injection in adult subjects with type 2 diabetes mellitus (T2DM) who have poor glycemic control after dietary exercise intervention only.

The proposed plan is to enroll 270 subjects with T2DM, using stratified block group randomization, with the stratification factor being baseline HbA1c (≤8.5% or >8.5%), and randomly assign them to the 1.2 mg JY09 injection group (n=90 subjects), the 2.4 mg JY09 injection group (n=90 subjects), and the placebo group (n=90 subjects) in a 1:1:1 ratio.

The trial was divided into 4 phases, i.e., a screening period of 2 weeks, a single-blind introduction period of 4 weeks, a treatment period of 54 weeks (26 weeks for the core treatment period and 28 weeks for the extended treatment period), and a safety follow-up period of 4 weeks. Total 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age and ≤75 years of age at the time of signing the informed consent form.
2. Those who meet the World Health Organization（WHO）1999 diagnostic criteria for type 2 diabetes mellitus and the WHO Recommendations for the Use of Glycosylated Haemoglobin (HbA1c) for Diagnosis (2011) supplemental diagnostic criteria for a diagnosis of T2DM for ≥ 12 weeks.
3. Those who received dietary and exercise interventions for ≥8 weeks prior to screening and who had not received any antidiabetic medications in the 8 weeks prior to screening.
4. HbA1c ≥7.5% and ≤11.0% at screening (local laboratory) and HbA1c ≥7.0% and ≤10.5% before randomization (V3) (central laboratory).
5. FPG 13.9 mmol/L at screening (local laboratory) and FPG 13.9 mmol/L before randomization (V3) (central laboratory).
6. Body mass index (BMI) ≥18.5 kg/m2 and ≤35.0 kg/m2 at screening and before randomization (V3).
7. Able to understand and willing to sign a written informed consent form (ICF) and comply with the study protocol.

Exclusion Criteria:

1. People diagnosed with type 1 diabetes or other types of diabetes.
2. Those who have used other hypoglycemic agents within 8 weeks prior to screening or prior to randomization (V4), or those who have used medications that may affect glucose metabolism, such as systemic glucocorticoids (except for inhalation or topical topical use), growth hormones, etc.
3. Acute complications of diabetes, such as diabetic ketoacidosis or hyperglycemic hyperosmolar state, within 6 months prior to screening or prior to randomization.
4. Severe chronic complications of diabetes mellitus (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within 6 months prior to screening, which are assessed by the investigator to be unsuitable for participation in this clinical study.
5. Persons who have had a severe trauma or serious infection within 1 month prior to screening or prior to randomization (V4) that may affect glycemic control, and persons who currently have a complicated or refractory urinary or genital tract infection.
6. Suffering from any condition at screening or prior to randomization (V4) that may cause hemolysis or red blood cell instability that would interfere with the measurement of HbA1c levels, such as hemolytic anemia.
7. Subjects who have abnormal thyroid function tests at Screening and require medication, or subjects who are being treated with thyroid-related medications whose thyroid function is still not well controlled at Screening.
8. Those with any of the following abnormalities on serologic testing at screening:

1）Positive human immunodeficiency virus antibodies or syphilis spirochete-specific antibodies; 2）Hepatitis C antibody positive; 3）Hepatitis B virus surface antigen (HBsAg) positive and hepatitis B viral load (HBV-DNA) above the lower limit of laboratory testing (HBV-DNA is added only if HBsAg is positive); 9. The subject has other conditions that, in the judgment of the investigator, make participation in this clinical study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, Week 26
  Change in glycated hemoglobin (HbA1c) values relative to baseline after 26 weeks of treatment.

SECONDARY OUTCOMES:
The proportion of HbA1c <6.5% and <7% | Baseline, Week 26,Week 54
  Proportion of subjects with HbA1c <7% and HbA1c <6.5% after 26 and 54 weeks of treatment.
HbA1c | Baseline, Week 6,Week 10,Week 14,Week 20,Week 38,Week 54
  Change in HbA1c relative to baseline after 6, 10, 14, 20, 38, and 54 weeks of treatment.
fasting plasma glucose (FPG) | Baseline, Week 6,Week 10,Week 14,Week 20,Week 38,Week 54
  Change in fasting plasma glucose (FPG) relative to baseline after 6, 10, 14, 20, 38, and 54 weeks of treatment.
fasting insulin | Baseline, Week 14,Week 26,Week 54
  Change in fasting insulin relative to baseline after 14, 26, and 54 weeks of treatment.
Homeostatic Model Assessment of Insulin Resistance(HOMA-IR) | Baseline,Week 26,Week 54
  Change in HOMA-IR relative to baseline after 26 and 54 weeks of treatment.
Health Survey Short Form (SF-36) | Baseline,Week 26,Week 54
  Value of change in Health Survey Short Form (SF-36) scores relative to baseline after 26 and 54 weeks of treatment.
blood pressure | Baseline,Week 26,Week 54
  Change in blood pressure (sitting) relative to baseline after 26 and 54 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No